CLINICAL TRIAL: NCT04060199
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled, Multi-center Study to Assess the Efficacy and Safety of Viltolarsen in Ambulant Boys With Duchenne Muscular Dystrophy (DMD)
Brief Title: Study to Assess the Efficacy and Safety of Viltolarsen in Ambulant Boys With DMD (RACER53)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NS Pharma, Inc. (Industry)
Collaborators: Nippon Shinyaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NS-065/NCNP-01-301
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — viltolarsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Viltolarsen (Experimental): Patients amenable to exon 53 skipping will receive viltolarsen intravenous (IV) infusions, weekly, at 80 mg/kg for up to 48 weeks.
  Interventions: Drug: Viltolarsen
- Placebo (Placebo Comparator): Patients amenable to exon 53 skipping will receive placebo intravenous (IV) infusions, weekly, for up to 48 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Viltolarsen — IV infusion
  Other Names: NS-065/NCNP-01
  Arms: Viltolarsen
Drug: Placebo — IV infusion
  Arms: Placebo

SUMMARY:
The main objective of this study is to evaluate the efficacy of Viltolarsen compared to placebo in Duchenne muscular dystrophy (DMD) patients amenable to exon 53 skipping.

DETAILED DESCRIPTION:
This is a Phase 3 randomized, double-blind, placebo-controlled, multi-center study to assess the efficacy and safety of Viltolarsen in ambulant boys with Duchenne muscular dystrophy. Eligible patients with out-of-frame deletion mutations amenable to exon 53 skipping will be randomized to receive once weekly intravenous (IV) infusions of 80 mg/kg Viltolarsen or placebo for up to 48 weeks.

The study will enroll approximately 74 patients amenable to exon 53 skipping. Clinical efficacy will be assessed at regularly scheduled study visits, including functional tests such as Time to Stand Test (TTSTAND), Time to Run/Walk 10 Meters Test (TTRW), Six-minute Walk Test (6MWT), North Star Ambulatory Assessment (NSAA), Time to Climb 4 Steps Test (TTCLIMB) and Hand-held dynamometer (elbow extension, elbow flexion, knee extension and knee flexion on the dominant side only).

Safety will be assessed through the collection of adverse events (AEs), laboratory tests, electrocardiograms (ECGs), vital signs, and physical examinations throughout the study.

Blood samples will be taken periodically throughout the study to assess the pharmacokinetics of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 4 years and < 8 years of age
* Confirmed DMD mutation(s) in the dystrophin gene that is amenable to skipping of exon 53 to restore the dystrophin mRNA reading frame
* Able to walk independently without assistive devices
* TTSTAND < 10 seconds
* Stable dose of glucocorticoid (GC) for at least 3 months prior to study entry and is expected to remain on stable dose of GC treatment for the duration of the study
* Other inclusion criteria may apply

Exclusion Criteria:

* Current or history of chronic systemic fungal or viral infections
* Acute illness within 4 weeks prior to the first dose of study drug
* Evidence of symptomatic cardiomyopathy (Note: Asymptomatic cardiac abnormality on investigation would not be exclusionary)
* Allergy or hypersensitivity to the study drug or to any of its constituents
* Severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the investigator
* Previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety, make it unlikely that treatment and follow-up will be correctly completed or impair the assessment of study results, in the opinion of the investigator;
* Surgery within the 3 months prior to the first dose of study drug or surgery is planned for anytime during the duration of the study
* Participant has positive test results for hepatitis B antigen, hepatitis C antibody or human immunodeficiency virus (HIV)
* Currently taking any other investigational drug or has taken any other investigational drug within 3 months prior to the first dose of study drug or within 5 times the half-life of a medication, whichever is longer
* Previously enrolled in an interventional study of viltolarsen
* Currently taking any other exon skipping agent or has taken any other exon skipping agent within 3 months prior to the first dose of study drug
* Having taken any gene therapy
* Other exclusion criteria may apply

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 77 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (2):
  - University of California Davis Medical Center, Sacramento, California
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
- Australia (3):
  - Queensland Children's Hospital, Brisbane
  - Perth Children's Hospital, Nedlands
  - The Childrens Hospital at Westmead, Westmead
- Canada (3):
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - Alberta Children's Hospital, Calgary
  - CHU de Quebec Research Centre, Québec
- Chile (2):
  - Hospital de Niños Roberto del Rio, Santiago
  - Pontificia Universidad Católica de Chile, Santiago
- China (5):
  - Chinese PLA General Hospital, Beijing
  - The Third Medical Center of PLA General Hospital, Beijing
  - Hunan Children's Hospital, Changsha
  - Children's Hospital of Fudan University, Shanghai
  - Shenzhen Children's Hospital, Shenzhen
- Greece (2):
  - Agia Sofia Children's Hospital, Athens
  - Hippokration General Hospital of Thessaloniki, Thessaloniki
- Hong Kong Children's Hospital, Kowloon Bay, Hong Kong
- Fondazione Policlinico Universitario A. Gemelli - Universita Cattolica del Sacro Cuore, Rome, Italy
- Mexico (2):
  - Hospital Angeles Chihuahua, Chihuahua City
  - Instituto Nacional de Pediatria, Mexico City
- Netherlands (2):
  - Radboud Universitair Medisch Centrum, Nijmegen, Gelderland
  - Leids Universitair Medisch Centrum, Leiden
- New Zealand Clinical Research Ltd, Auckland, New Zealand
- Rikshospitalet, Oslo, Norway
- Russia (3):
  - Russian National Research Medical University n.a. N.I.Pirogov, structural branch - Research Clinical Institute of Pediatrics n.a. Academician Yu. E. Veltishchev, Moscow
  - "Saint Petersburg State Paediatric Medical University" based at Consultative and Diagnostic Centre, Saint Petersburg
  - Tomsk National Research Medical Center of Russian Academy of Sciences, Tomsk
- South Korea (2):
  - Pusan National University Yangsan Hospital, Pusan
  - Seoul National University Hospital, Seoul
- Spain (2):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitario La Paz, Madrid
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
- Yeditepe University Kosuyolu Hospital, Istanbul, Turkey (Türkiye)
- State Institution "Ukrainian Medical rehabilitation Center for Children with organic disorders of the nervous system of the Ministry of Health of Ukraine", Kyiv, Ukraine
- United Kingdom (4):
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Hospital for Children - Glasgow, Glasgow
  - University College London Institute of Child Health, London
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study from April 14, 2020 to October 19, 2023 at 30 sites in 17 countries, predominantly in Europe, Asia, North America, and South America
Pre-assignment Details: Eighty-three patients were screened. Six patients were screen failed due to failure to satisfy inclusion/exclusion criteria. Analysis Populations for all randomized patients was 77 patients.
Period: Overall Study
Arm/Group | Viltolarsen | Placebo
Started | 38 | 39
Completed | 36 | 38
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: The ITT Population was defined as all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Viltolarsen | Placebo | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.5 (1.20) | 5.7 (1.16) | 5.6 (1.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 38 | 39 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 36 | 33 | 69
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 11 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 26 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Weight [Mean (Standard Deviation); unit: kg] | 21.12 (4.354) | 20.70 (4.277) | 20.91 (4.292)
Height [Mean (Standard Deviation); unit: cm] | 110.9 (9.78) | 111.8 (7.78) | 111.4 (8.78)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 17.053 (1.9427) | 16.439 (2.1105) | 16.742 (2.0396)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Time to Stand (TTSTAND) Velocity
Description: The change from baseline for velocity converted from TTSTAND was compared between the viltolarsen-treated patients and the placebo-treated patients. TTSTAND was assessed as the time it takes the participant to go from lying flat on the floor to standing. The time measured for TTSTAND was converted to a velocity expressed as rise per second.
Time Frame: baseline, Week 13, 25, 37, 49
Population: The modified ITT (mITT) Population was set as the analysis population. The mITT Population was defined as all randomized patients who received at least 1 dose of IP and had a baseline assessment and at least 1 post baseline efficacy assessment. The change from baseline for velocity converted from TTSTAND was compared between the viltolarsen-treated patients and the placebo-treated patients using a mixed-effect model for repeated measures (MMRM) analysis.
Measure: Least Squares Mean (Standard Error); unit: rise/s
Arm/Group | Viltolarsen | Placebo
Number analyzed (Participants) | 37 | 38
rise/s
  Week 13 | 0.026 (0.0103) | 0.013 (0.0104)
  Week 25: number analyzed (Participants) | 36 | 38
  Week 25 | 0.027 (0.0100) | 0.014 (0.0100)
  Week 37: number analyzed (Participants) | 35 | 36
  Week 37 | 0.027 (0.0107) | 0.027 (0.0108)
  Week 49: number analyzed (Participants) | 33 | 35
  Week 49 | 0.009 (0.0096) | 0.013 (0.0096)

ADVERSE EVENTS:
Time Frame: Up to 48 weeks
Description: Incidence of Adverse Events as assessed by CTCAE v4.03
Arm/Group | Viltolarsen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 2/38 | 3/39
Other Adverse Events (participants affected / at risk) | 33/38 | 37/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viltolarsen (N=38) | Placebo (N=39)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viltolarsen (N=38) | Placebo (N=39)
COVID-19 (Infections and infestations) | 12 (13) | 12 (13)
Upper respiratory tract infection (Infections and infestations) | 10 (18) | 9 (12)
Nasopharyngitis (Infections and infestations) | 9 (25) | 7 (16)
Rhinitis (Infections and infestations) | 6 (10) | 3 (5)
Gastroenteritis (Infections and infestations) | 3 (4) | 4 (4)
Influenza (Infections and infestations) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (3) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Hordeolum (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (3)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2)
Varicella (Infections and infestations) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 10 (12) | 13 (19)
Fatigue (General disorders) | 3 (3) | 1 (1)
Influenza-like illness (General disorders) | 2 (2) | 2 (3)
Administration site extravasation (General disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 7 (13)
Vomiting (Gastrointestinal disorders) | 4 (4) | 11 (12)
Abdominal pain (Gastrointestinal disorders) | 4 (10) | 6 (11)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Feces soft (Gastrointestinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 5 (7)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Blood triglycerides increased (Investigations) | 3 (4) | 2 (2)
Protein urine present (Investigations) | 2 (3) | 3 (5)
Blood cholesterol increased (Investigations) | 1 (2) | 2 (2)
Urine protein:creatinine ratio increased (Investigations) | 2 (3) | 1 (1)
Beta 2 microglobulin urine increased (Investigations) | 0 (0) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2)
Crystal urine present (Investigations) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 5 (6) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2) | 2 (3)
Urine abnormality (Renal and urinary disorders) | 3 (4) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Headache (Nervous system disorders) | 3 (3) | 5 (8)
Tachycardia (Cardiac disorders) | 3 (3) | 2 (2)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 3 (4) | 1 (3)
Hematoma (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The most restrictive relevant agreement on the PI provides that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is not less than 30 days from the time submitted to the sponsor for review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT04060199/Prot_SAP_000.pdf